CLINICAL TRIAL: NCT06288997
Title: TACS Intervention for Methamphetamine Addiction
Acronym: tACS for MUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFYuan_tACS
Record Dates: First submitted 2023-11-21; First posted 2024-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Methamphetamine Use Disorder
Keywords: transcranial alternating current stimulation; Methamphetamine use disorder; craving

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tACS group (Active Comparator): In the active group, the intervention is carried out using Hi-tACS with an intensive current of 15mA and a frequency of 77.5 Hz. Each intervention session lasts for 40 minutes, with two sessions conducted daily - one in the morning and one in the afternoon. The intervention is spread over a 10-day period, with sessions taking place five days per week, totaling two weeks.
  Interventions: Device: Active transcranial alternating current stimulation
- Sham tACS group (Sham Comparator): The sham group undergoes sessions with the same technical settings, designed to produce similar scalp sensations but without effective penetration of the electric field into the brain. Each session lasts for 40 minutes, with two sessions conducted daily - one in the morning and one in the afternoon. The intervention is spread over a 10-day period, with sessions taking place five days per week, totaling two weeks.
  Interventions: Device: Sham transcranial alternating current stimulation

INTERVENTIONS:
Device: Active transcranial alternating current stimulation — Hi-tACS with a current level of 15mA with a patented frequency of 77.5Hz.
  Arms: Active tACS group
Device: Sham transcranial alternating current stimulation — The device for the sham group has the same appearance and technical settings as the one used in the active group, designed to produce similar sensations on the scalp, but without effective penetration of the electric field into the brain.
  Arms: Sham tACS group

SUMMARY:
In 2021, nearly 296 million people worldwide used psychoactive substances, highlighting a significant need for effective interventions for disorders such as Methamphetamine Use Disorder (MUD). Despite existing treatments, including behavioral therapies and medications, the relapse rates remain high, signaling the need for more potent and targeted approaches. This clinical trial investigates high-intensity transcranial alternating current stimulation (Hi-tACS), a non-invasive method that applies 15mA electrical currents with a patented frequency of 77.5Hz to modulate brain activity. Hi-tACS has shown promise in preliminary studies for its ability to reduce drug cravings significantly by influencing brain regions crucial in addiction. The primary aim of this study is to evaluate the effectiveness of Hi-tACS in curbing cravings in individuals with MUD. As secondary objectives, the trial will also explore the potential benefits of Hi-tACS in alleviating other clinical symptoms, enhancing cognitive performance, and positively influencing brain activity. This study seeks to establish Hi-tACS as a more effective treatment option that could lead to substantially lower relapse rates for individuals with MUD.

DETAILED DESCRIPTION:
The study will be conducted at multiple drug rehabilitation centers in China. The procedure includes screening, pre-intervention evaluation (baseline), a 2-week intervention (twice daily sessions, 40 minutes each, totaling 20 sessions), post-intervention evaluation, and follow-up evaluations at 2 weeks and 3 months.

During the screening phase, participants are recruited and undergo a health interview to determine eligibility. If eligible, participants sign informed consent and are randomly assigned to one of two groups (active or sham).

At baseline, participants report demographic information and complete various questionnaires, cognitive tasks, and electroencephalogram (EEG) recordings to assess craving, clinical symptoms, and cognitive abilities.

During the intervention phase, tACS stimulates the scalp with three Nexalin electrodes (Nexalin Technology, Inc., Houston, TX, USA): electrodes are placed according to the international 10/20 system for EEG recording. A 4.45 × 9.53 cm electrode is placed above the forehead (Fpz, Fp1, and Fp2), and two 3.18 × 3.81 cm electrodes are placed above both mastoid areas. The active group receives 77.5 Hz tACS for 40 minutes per session. The sham group receives treatment with identical technical parameters, which induce scalp sensations but without penetration of the electric field into the brain. After each session, any side effects reported by participants are recorded to ensure safety and feasibility.

Post-intervention evaluation, as well as the 2-week and 3-month follow-up evaluations, mirror the pre-intervention assessments.

Sample size was calculated using GPower 3.1.9.4. Since Hi-tACS has not been previously investigated in drug addiction, an effect size of 0.15 was chosen. The power is set at 80%, and a two-tailed significance level is maintained at 5%. The calculations suggest a total sample size of 62. Considering potential dropout during treatment, the sample size was set at 70 (35 per group).

Throughout the intervention, patients, operators, and raters remain blinded to treatment conditions. To ensure study quality, researchers and drug rehabilitation staff will collaborate throughout the process, and data will be converted to electronic versions after each evaluation.

ELIGIBILITY:
The inclusion criteria include:

1. ages between 18 and 70;
2. education level of at least primary school;
3. confirmed diagnosis of MUD as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
4. a subjective craving score of 30 or higher;
5. absence of any other behavioral, pharmacological, or physical treatments during the trial.

The exclusion criteria include:

1. significant neurological or serious psychiatric disorders;
2. concurrent substance use disorders;
3. previous treatments with electroconvulsive therapy, transcranial magnetic stimulation, or transcranial direct current stimulation;
4. presence of a cochlear implant, cardiac pacemaker, implanted neurological device, or cerebral metal;
5. current pregnancy or lactation;
6. severe withdrawal symptoms;
7. engagement in other clinical studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective craving | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Subjective craving is measured by using Analogue Scale (VAS) for craving after watching video stimulus, ranging from 0 to 100, where 0 indicates no craving at all and 100 represents an extremely intense craving.
Objective craving | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Objective craving is measured by using the EEG recording to reflect the brain activity of individuals to the drug-related videos and pictures. EEG data were recorded when participants watch videos in Video-induced Craving Task (VCT) and when participants see pictures in Picture-induced Craving Task (PCT). The amplitude of late positive potential (LPP) was considered as a major outcome of the drug-cue related ERP, higher LPP is related to higher craving.

SECONDARY OUTCOMES:
Resting-state brain activity | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  based on resting-state EEG, the five power oscillations will be calculated (Delta band, Theta band, Alpha band, Beta band, and Gamma band).
Depression status | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  The depression status is measured by Beck Depression inventory scale. The questionnaire is a 21-question multiple-choice self-report inventory, score ranged from 0 to 63, high score means worse depression.
Anxiety status | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Anxiety status is measured by Beck anxiety inventory scale,it consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63). higher score means worse anxiety.
Sleep status | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Sleep status measured by Pittsburgh Sleep Quality Index scale (PSQI). The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Impulsivity | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Impulsivity is measured by Barratt Impulsiveness Scale, the total scores can range from 30 to 120. Higher score means higher impulsivity.
Uncertainty decision-making | The day before intervention, the day after intervention, 2 weeks after intervention and 3 months after intervention.
  Uncertainty decision-making ability is measured by using choice under risk and ambiguity. The score of probability for uncertainty choice is the major outcome, higher means more inclined to take risks. ERP (event-related potential) is also analyzed during decision-making. Higher amplitude of ERP means more inclined to take risks.

OTHER OUTCOMES:
side effect measurements | every day after each intervention time for the 2 weeks intervention time period
  The side effect is measured by Side effect scale, including ten types of adverse effects, such as headache, pricking, sleeplessness etc. The score ranged from 0 to 100, higher score indicates severe adverse effect.

CONTACTS AND LOCATIONS:
Overall Officials: Ti-fei Yuan, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (5):
- China (5):
  - Beijing Tiantanghe Addiction Rehab Center, Beijing, Beijing Municipality
  - Hubei Shizishan Drug Rehabilitation Center, Wuhan, Hubei
  - Da Lian Shan Institute of Addiction Rehabilitation, Nanjing, Jiangsu
  - Tai Hu Institute of Addiction Rehabilitation, Suzhou, Jiangsu
  - Sichuan Drug Rehabilitation Center, Deyang, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
share all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within twelve months after the trial complete
Access Criteria: share to health care personnel, patients and the general public.
URL: http://clinicaltrials.gov